CLINICAL TRIAL: NCT00584558
Title: Long-Term Follow-Up of Catheter Ablation
Brief Title: Long-Term Follow-Up of Patients Undergoing Catheter Ablation
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Karen Beckman, MD, Principal Investigator, University of Oklahoma
Other Study IDs: 1239
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-05

CONDITIONS: Arrhythmia
Keywords: Arrhythmia; Catheter Ablation
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients undergoing catheter ablation.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — Catheter Ablation of arrhythmias
  Other Names: All approved ablation catheters; Investigational ablation catheters

SUMMARY:
The purpose of this study is to assess the long-term effects of catheter ablation procedures performed at the OU Medical Center.

DETAILED DESCRIPTION:
The purpose of this study is to assess the long-term effects of catheter ablation procedures performed at this institution, including recurrence of the ablated arrhythmia and any late complications.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing catheter ablation at the OU Medical Center

Exclusion Criteria:

* Prisoners
* Refusal to participate

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing catheter ablation at the OU Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 2420 (Actual)
Dates: Start 2001-02; Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Beckman, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-Catheter Ablation: There is only one arm. Observational study of patients between the ages of 1 and 100 years undergoing catheter ablation of arrhythmias at OUHSC using FDA approved devices. No investigational devices in this study.
Period: Overall Study
Arm/Group | 1-Catheter Ablation
Started | 2420
Completed | 2420
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Observational Arm: All patients studied
Arm/Group | Observational Arm
Number analyzed (Participants) | 2420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 678
  Between 18 and 65 years | 1306
  >=65 years | 436
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 992
  Male | 1428
Region of Enrollment [Number; unit: participants]
  United States | 2420

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Arrhythmia Recurrence
Description: Number and % patients with documented arrhythmias recurrences
Time Frame: 0-10 years
Population: Patients who underwent ablation of arrhythmias
Measure: Count of Participants; unit: Participants
Arm/Group | 1-Catheter Ablation
Number analyzed (Participants) | 2420
Participants | 100

2. Secondary Outcome: Number of Patients With Complications From Catheter Ablation
Description: Number and % of patients with major adverse events as recorded in the medical record
Time Frame: 0-10 years
Measure: Count of Participants; unit: Participants
Groups:
- 1-Observational: There is only one arm. Observational study of patients between the ages of 1 and 100 years undergoing catheter ablation of arrhythmias at OUHSC using FDA approved devices. No investigational devices in this study.
Arm/Group | 1-Observational
Number analyzed (Participants) | 2430
Participants | 72

ADVERSE EVENTS:
Groups:
- Observational Arm: Patients undergoing catheter ablation.
  Catheter Ablation: Catheter Ablation of arrhythmias
Arm/Group | Observational Arm
All-Cause Mortality (participants affected / at risk) | 6/2420
Serious Adverse Events (participants affected / at risk) | 72/2420
Other Adverse Events (participants affected / at risk) | 24/2420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Arm (N=2420)
Cardiac Tamponade (Cardiac disorders) | 72 (72) — Cardiac Tamponade 3%
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Arm (N=2420)
IVC thrombus (Vascular disorders) | 24 (24) — IVC thrombus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No